CLINICAL TRIAL: NCT00151268
Title: Genotype - Phenotype Correlations of Late Infantile Neuronal Ceroid Lipofuscinosis
Brief Title: Genotype - Phenotype Correlations of LINCL
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Nathan's Battle Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 0401007011
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Batten Disease; Late-Infantile Neuronal Ceroid Lipfuscinosis
Keywords: Batten Disease; Late Infantile Neuronal Lipofuscinosis; LINCL
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In a separate protocol the Department of Genetic Medicine is proposing to carry out a study using gene transfer to treat the central nervous system (CNS) manifestations of late infantile neuronal ceroid lipofuscinosis (LINCL), a fatal, rare, recessive disorder of the (CNS) in children. In the context that there is little known about the genotype - phenotype correlations of LINCL, and that our referral far exceed the number (n=11) of children that will be entered into the gene transfer protocol, we are proposing to capitalize on this unique opportunity to evaluate this disorder in this separate study. In this context, the aim of this protocol is to study the genotype - phenotype correlations of the CNS manifestations of late infantile neuronal ceroid lipofuscinosis. This will be accomplished by comparing the genotype to a neurologic assessment, and LINCL clinical rating scale; magnetic resonance imaging (MRI) and magnetic resonance spectroscopic (MRS) assessments of the CNS; and routine clinical evaluations.

DETAILED DESCRIPTION:
This proposed clinical protocol is designed to assess genotype - phenotype correlations of LINCL, including a preliminary assessment regarding the genotype - phenotype correlations of progressive CNS deterioration inherent to this disorder. The trial will include the primary endpoint of neurological assessment including the LINCL clinical rating scale and parental evaluations; and the secondary endpoint of magnetic resonance imaging (MRI) and magnetic resonance spectroscopic (MRS) assessments of the CNS.

The study will be carried out in children diagnosed with LINCL in all stages. The staging is based on a modification of the scale of Steinfeld et al (Steinfeld, 2002). The study anticipates a total n=30 children assessed over a period of 18 months. Of these, we anticipate that approximately two-thirds will not be entered into the proposed gene therapy protocol and thus approximately n=20 will be available for this study to be reassessed at 1 year. Thus, we anticipate that we will be able to capture a one-time genotype - phenotype snapshot for all n=30, and a 1 year genotype - phenotype progression assessment for n=20.

ELIGIBILITY:
Inclusion Criteria:

* A definitive diagnosis of late infantile neuronal ceroid lipofuscinosis
* Between the age of 2 and 18 years
* Not previously participated in a gene transfer study for LINCL.
* Parents of study participants must agree to comply in good faith with the conditions of the study, including attending all of the required baseline and follow-up assessments.
* Both parents or legal guardians must give consent for their child's participation in the research study.

Exclusion Criteria:

* Individuals with heart disease that would be a risk for anesthesia.
* Concurrent participation in any other FDA approved Investigational New Drug clinical protocol is not allowed, although the Principal Investigator will work with other doctors to accommodate specific requests (e.g., a study of nutritional supplements probably would not be a disqualification).
* Individuals who have a contraindication to MRI/MRS assessment including: (1) heart pacemaker and/or related implants; (2) metal fragment/chip in the eye or other sites; (3) an aneurysm clip in their brain; and (4) metallic inner ear implants.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will be carried out in children diagnosed with LINCL in all stages.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2004-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Correlation analysis between genotype (genetic constitution) and baseline | 18 months

SECONDARY OUTCOMES:
Correlation analysis between genotype and rate of CNS decline | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G. Crystal, MD, Principal Investigator — Weill Medical College of Cornell University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sondhi D, Kaminsky SM, Rosenberg JB, Rostami MR, Hackett NR, Crystal RG. Twenty-Year Survival Analysis of Adeno-Associated Virus Vector Serotype 2-Mediated Gene Therapy to the Central Nervous System for CLN2 Disease. Hum Gene Ther. 2024 Jan;36(1-2):28-35. doi: 10.1089/hum.2024.182. Epub 2025 Jan 2. PMID 39745261
- [Derived] Worgall S, Sondhi D, Hackett NR, Kosofsky B, Kekatpure MV, Neyzi N, Dyke JP, Ballon D, Heier L, Greenwald BM, Christos P, Mazumdar M, Souweidane MM, Kaplitt MG, Crystal RG. Treatment of late infantile neuronal ceroid lipofuscinosis by CNS administration of a serotype 2 adeno-associated virus expressing CLN2 cDNA. Hum Gene Ther. 2008 May;19(5):463-74. doi: 10.1089/hum.2008.022. PMID 18473686
- [Derived] Worgall S, Kekatpure MV, Heier L, Ballon D, Dyke JP, Shungu D, Mao X, Kosofsky B, Kaplitt MG, Souweidane MM, Sondhi D, Hackett NR, Hollmann C, Crystal RG. Neurological deterioration in late infantile neuronal ceroid lipofuscinosis. Neurology. 2007 Aug 7;69(6):521-35. doi: 10.1212/01.wnl.0000267885.47092.40. PMID 17679671